CLINICAL TRIAL: NCT04195035
Title: Comparison of Air QTM Intubating Airway Versus Ambu-Aura Intubating Laryngeal Mask Obese Patients Under General Anaesthesia.
Brief Title: Comparison of Air QTM Intubating Airway Versus Ambu-Aura Intubating Laryngeal Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-19-2019
Record Dates: First submitted 2019-12-07; First posted 2019-12-11 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Airway Management; Obesity
Keywords: obesity; Air QTM intubating airway; Ambu-Aura intubating laryngeal mask
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air-Q intubating laryngeal airway mask (Experimental): Where Air-Q intubating laryngeal airway will be used for ventilation & intubation through fiberoptic bronchoscope.
  After complete muscle relaxation a suitable sized (according to the patient's weight and BMI) Air-Q will be lubricated inserted and the ventilator circuit will be connected to the device to ventilate the patient. The ventilator will be set with tidal volume 4-6 ml/kg at a respiratory rate 12-15 breath/minute to keep normocapnia (ETCO2=30-35 mmHg). Vitals (HR, ABP and O2 saturation) and ET CO2were recorded 5 minutes after device insertion.
  Then intubation using the fiberoptic bronchoscope will be started through the supraglottic device, laryngeal view grade will be recorded, success of endotracheal intubation through the device and time of intubation (time starting from disconnection of the circuit from the device to use the fiberoptic brochoscope for intubation till tube insertion in the trachea).
  Interventions: Device: Air-Q intubating laryngeal airway
- Ambu-Aura intubating laryngeal mask (Experimental): Ambu-Aura intubating laryngeal mask will be used for ventilation & intubation through fiberoptic bronchscope.
  After complete muscle relaxation a suitable sized (according to the patient's weight and BMI) Ambu-Aura laryngeal mask will be lubricated inserted and the ventilator circuit will be connected to the device to ventilate the patient. The ventilator will be set with tidal volume 4-6 ml/kg at a respiratory rate 12-15 breath/minute to keep normocapnia (ETCO2=30-35 mmHg). Vitals (HR, ABP and O2 saturation) and ET CO2 will be recorded 5 minutes after device insertion.
  Then intubation using the fiberoptic bronchoscope will be started through the supraglottic device, laryngeal view grade will be recorded, success of endotracheal intubation through the device and time of intubation (time starting from disconnection of the circuit from the device to use the fiberoptic brochoscope for intubation till tube insertion in the trachea).
  Interventions: Device: Ambu-Aura intubating laryngeal mask

INTERVENTIONS:
Device: Air-Q intubating laryngeal airway — Air-Q intubating laryngeal airway will be used for ventilation & intubation through fiberoptic bronchoscope.
  Arms: Air-Q intubating laryngeal airway mask
Device: Ambu-Aura intubating laryngeal mask — Ambu-Aura intubating laryngeal mask will be used for ventilation & intubation through fiberoptic bronchscope.
  Arms: Ambu-Aura intubating laryngeal mask

SUMMARY:
Supraglottic airway devices are important tools for airway management. Supraglottic airway devices have been introduced into brief surgical interventions because they are less invasive than intubation and safer than mask to maintain the patency of airway after induction of anesthesia. They are inserted via the oral route and can be used in emergency conditions when tracheal intubation and mask anesthesia are challenging.

Air Q intubating airway and Ambu Aura intubating laryngeal mask are two Supraglottic airway devices that are widely used.

Aim of the work is to compare Air-Q intubating laryngeal airway versus Ambu-Aura intubating laryngeal mask regarding sealing pressure and Fiberoptic intubation in class II obese patients.

DETAILED DESCRIPTION:
Randomized comparative trial that will be performed in Kasr Al Ainy hospital, Cairo University, Cairo, Egypt.ASA II patients from 20 to 50 years of age, undergoing minor surgry were included in this study. 40 patients will be allocated into 2 equal groups using computerized software and enclosed in sealed opaque envelopes:

GQ ( n=20 ): Where Air-Q intubating laryngeal airway will be used for ventilation & intubation through fiberoptic bronchoscope.

GA ( n=20 ): Where Ambu-Aura intubating laryngeal mask will be used for ventilation & intubation through fiberoptic bronchscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years old.
* Sex: both genders.
* With American society of anaesthesiologists (ASA) physical activity II.
* Scheduled for elective surgery under general anaesthesia requiring endotracheal tube.
* Class II obese patients (BMI 34.9 - 39.9 kg/m2).
* Surgery: short time procedures ≥ 60 minutes, ≤ 120 minutes e.g.: breast surgery, elbow or foot surgery.

Exclusion Criteria:

* • Patient refusal.

  * Patients with any respiratory tract abnormalities as laryngeal masses & facial deformities as fracture mandible.
  * Patients with risk of pulmonary aspiration as in full stomach patients.
  * Patients at risk of regurgitation of gastric content as in gastroesophageal reflux disease (GERD) and pregnant females.
  * Emergency operation.
  * Patients with obstructive sleep apnea.
  * Patients prepared for laparotomy or laparoscopic procedures.
  * Patients with risk of bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-01-10 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
airway seal pressure | 1 minute
  Measuring the seal pressure above which the oropharyngeal leak through the supraglottic device will occur (1 minute after confirmation of successful insertion).

SECONDARY OUTCOMES:
Success rate | 1 minute
  Success rate of device insertion
arterial blood pressure | 2 hours
  systolic and diastolic arterial blood pressure. • Stress response related to the device used.
heart rate | 2 hours
  • Stress response related to the device used
Laryngeal view grade. | 1 minute
  Grade 1: only larynx was seen, Grade 2: larynx plus the posterior surface of epiglottis were seen. Grade 3: larynx and anterior tip of epiglottis were seen with <50% visual obstruction of larynx.
  Grade 4: epiglottis down folded and its anterior surface were seen with >50% visual field obstruction.
  Grade 5: complete down folding of epiglottis and the larynx could not be seen directly
Success rate of intubation by fiberoptic bronchoscope | 1 minute
  The success of the ventilation will be determined based on visible chest expansion, adequate tidal volume and drawing of 6 successive ETCO2 waves.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Lee JH, Han SW, Im YJ, Kang HJ, Lee JR. A randomized comparison of the i-gel with the self-pressurized air-Q intubating laryngeal airway in children. Paediatr Anaesth. 2015 Apr;25(4):405-12. doi: 10.1111/pan.12609. Epub 2015 Jan 6. PMID 25559870
- [Background] Jagannathan N, Kozlowski RJ, Sohn LE, Langen KE, Roth AG, Mukherji II, Kho MF, Suresh S. A clinical evaluation of the intubating laryngeal airway as a conduit for tracheal intubation in children. Anesth Analg. 2011 Jan;112(1):176-82. doi: 10.1213/ANE.0b013e3181fe0408. Epub 2010 Nov 16. PMID 21081777
- [Background] Yahaya Z, Teoh WH, Dintan NA, Agrawal R. The AMBU(R) Aura-i Laryngeal Mask and LMA Supreme: A Randomized Trial of Clinical Performance and Fibreoptic Positioning in Unparalysed, Anaesthetised Patients by Novices. Anesthesiol Res Pract. 2016;2016:4717061. doi: 10.1155/2016/4717061. Epub 2016 Oct 25. PMID 27847515
- [Background] Galgon RE, Schroeder KM, Han S, Andrei A, Joffe AM. The air-Q((R)) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. doi: 10.1111/j.1365-2044.2011.06863.x. Epub 2011 Aug 22. PMID 21880031